CLINICAL TRIAL: NCT01746810
Title: IR-guided Ablation (IRGA) Combined With Stereotactic Ablative Radiation (SABR) for Lung Tumors Larger Than 3 cm: Phase I Dose Escalation and Pilot Study With Companion Biomarker Analysis
Brief Title: IR-guided Ablation (IRGA) Combined With Stereotactic Ablative Radiation (SABR) for Large Lung Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Closed study as requested by PI due to lack of accruals
Sponsor: New Mexico Cancer Research Alliance (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INST 1206
Record Dates: First submitted 2012-11-26; First posted 2012-12-11 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Recurrent Non-small Cell Lung Cancer
Keywords: Metastatic; Lung Cancer; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis; Lung Neoplasms | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stereotactic Body RT and IRGA (Experimental): Patients undergo stereotactic body radiation therapy QD for a total of 5 fractions and then undergo IRGA (either radiofrequency ablation or microwave ablation) 1 week later.
  Interventions: Radiation: Stereotactic body RT and IRGA

INTERVENTIONS:
Radiation: Stereotactic body RT and IRGA — SABR Treatment with Dose escalation: Group 1: 40 Gy/5 fractions Group 2: 45 Gy/5 fractions Group 3: 50 Gy/5 fractions then IRGA procedure 1 week later with repeat lung biopsies, serum studies
  Other Names: Radiofrequency ablation; Microwave ablation

SUMMARY:
This phase I trial studies the side effects and best dose of stereotactic body radiation therapy when given together with ablation therapy in treating patients with non-small cell lung cancer or lung metastases. Ablation therapy, such as radiofrequency ablation uses a high-frequency, electric current to kill tumor cells. Ablation therapy, such as microwave ablation kills tumor cells by heating them to several degrees above normal body temperature. Stereotactic body radiation therapy may be able to send x-rays directly to the tumor and cause less damage to normal tissue. Giving ablation therapy together with stereotactic body radiation therapy may kill more tumor cells.

DETAILED DESCRIPTION:
This is a dose-escalation study of stereotactic body radiation therapy.

Patients undergo stereotactic body radiation therapy once daily (QD) for a total of 5 fractions and then undergo IRGA (either radiofrequency ablation or microwave ablation) 1 week later.

After completion of study treatment, patients are followed up at 4 weeks, every 3 months for 1 year, every 4 months for 1 year, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Pathological (histologically or cytologically) diagnosis of non-small cell lung cancer (NSCLC); or if lung tumor is considered to be metastases (even from primary NSCLC), then clinical diagnosis is sufficient
* For NSCLC: Staging workup at initial diagnosis demonstrates T2-T4N0M0, or T2-T4,N1-3,M1; node-positive patients will be allowed on study only if they have M1 disease; clinical diagnosis of M1 disease is sufficient
* Patient is deemed (a) to be medically inoperable after evaluation by thoracic surgeon based on, but not limited to the following: baseline forced expiratory volume in one second (FEV1) < 40% predicted, post-operative FEV1 < 30% predicted, severely reduced diffusion capacity, baseline hypoxemia/hypercapnia, coronary artery disease, end-organ damage, or (b): patient has refused surgery after thoracic surgery consultation
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* NSCLC only: pleural effusion, if present, will undergo routine assessment for malignancy; inability to obtain fluid or non-diagnostic cytology will not preclude eligibility
* Negative serum or urine pregnancy test within 4 weeks prior to registration in women with childbearing potential
* Able to provide written, informed consent
* Minimum of 4 weeks from last dose of chemotherapy to start of treatment

Exclusion Criteria:

* For NSCLC only: prior invasive malignancy (except non-melanoma skin cancer) unless disease-free for a minimum of 2 years, including previous history of lung cancer
* Prior radiation to the region of current cancer that would result in > 50% overlap of the old treatment field on the new treatment area based on radiation oncologist evaluation
* International normalization ratio (INR) of > 1.5
* Platelets of < 50,000 /uL
* Inability to meet maximum point dose constraints

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2015-10-13 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 30 to 90 days
  The MTD will be defined as the highest dose level where less than or equal to 33% patients incurred a dose-limiting toxicity (DLT). A DLT will be defined as an acute (within 30 days) or subacute (31-90 days) irreversible grade 3 or any grade 4-5 toxicity (using National Cancer Institute [NCI]-Common Toxicity Criteria [CTC] version 4.0 criteria) that is possibly, probably, and definitely attributed to the therapy.

SECONDARY OUTCOMES:
Survival | Up to 6 years
  Rates of local control, disease-free survival, and overall survival
Biomarker testing | 2 weeks
  Size of tissue samples sufficient for DNA analyses
Pathological Response | Up to 6 years
  Pathological response, changes in protein expression, and biomarker correlations with clinical outcome
Quality of Life | Up to 6 years
  Quality of life (European Organization for the Research and Treatment of Cancer [EORTC])

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Schroeder, MD, Principal Investigator — UNM Cancer Center
Locations (1):
- University of New Mexico Cancer Center, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: UNM Cancer Center — http://www.cancer.unm.edu
- See also: New Mexico Cancer Care Alliance — http://www.nmcca.org